CLINICAL TRIAL: NCT02719379
Title: Immune Response to Pneumococcal Polysaccharide Vaccine (23-valent) Predicts Asthma Status and Outcomes in Late Adolescents With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rohit Divekar (Other)
Responsible Party: Sponsor-Investigator, Rohit Divekar, Assistant Professor of Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15-005581
Record Dates: First submitted 2016-03-14; First posted 2016-03-25 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Asthmatics (Experimental): 19-20 year old asthmatics who agree to participate in study will have serum collected for analysis. PPSV23 vaccine [Pneumonococcal Polysaccharide Vaccine 23-valent (PPSV-23)] will be offered per the ACIP/CDC guidelines. Those who agree to receive the vaccine will have a second draw for serum 4-6 weeks post vaccination for immunization response. They will also be follow up after 1 year to assess for asthma control and outcomes. This arm will additionally allow for comparison of asthma outcomes and vaccine response
  Interventions: Biological: Pneumonococcal Polysaccharide Vaccine 23-valent (PPSV-23)
- Non-asthmatics (Active Comparator): 19-20 year old non-asthmatic smokers who agree to participate in study will have serum collected for analysis. PPSV23 vaccine [Pneumonococcal Polysaccharide Vaccine 23-valent (PPSV-23)] will be offered per the ACIP/CDC guidelines. Those who agree to receive the vaccine will have a second draw for serum 4-6 weeks post vaccination for immunization response. This arm will allow for comparison of vaccine response between asthmatics and non-asthmatics (smokers)
  Interventions: Biological: Pneumonococcal Polysaccharide Vaccine 23-valent (PPSV-23)
- Asthmatics - Serum Stored (Other): Once the accrual for the experimental arm is met, 19-20 year old asthmatics who wish to participate in study will have serum collected for analysis. PPSV23 vaccine [Pneumonococcal Polysaccharide Vaccine 23-valent (PPSV-23)] will be offered per the ACIP/CDC guidelines. This arm will allow for study of baseline vaccine titers to pneumococcus in asthmatics at same time increase the vaccine uptake in the community.
  Interventions: Biological: Pneumonococcal Polysaccharide Vaccine 23-valent (PPSV-23)

INTERVENTIONS:
Biological: Pneumonococcal Polysaccharide Vaccine 23-valent (PPSV-23)
  Other Names: Pneumovax

SUMMARY:
Advisory Committee for Immunization Practices (ACIP) from the Centers for Disease Control (CDC) recommends that children (6-18 years) and adults (≥19 years old) with chronic lung condition such as asthma or cigarette smoking be vaccinated with Pneumococcal vaccine (PPSV23). The purpose of this study is to increase awareness of vaccination to late adolescents with asthma and smokers (social aspect of study), and to recommend vaccination (which is the clinical aspect). Individuals who agree to receiving vaccine will be enrolled in research to determine whether late adolescents with and without asthma (smokers) have distinctive pneumococcal vaccine response patterns and whether such patterns are associated with subsequent variance in asthma outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Reside in Olmsted County, Minnesota (defined by Olmsted County address in medical record within one year prior to last follow-up date as of data abstraction)
* Receive medical care from Mayo Clinic clinical practice
* Signed research authorization for using medical record for research

Exclusion Criteria:

* Diagnosis of an immunodeficiency (primary and secondary)
* Previous or current diagnosis of a Rheumatological disorders (Rheumatoid arthritis, Lupus, Sjögren, and vasculitis), cancer (chronic lymphocytic leukemia, non-Hodgkin lymphoma, and B-cell malignancy), diabetes, active infection (pneumonia, otitis media, HIV, and EBV), other chronic diseases (multiple sclerosis, etc), renal disease such nephritic syndrome, and protein losing enteropathy
* Current or previous use (within the last 6 months) of systemic corticosteroids, and other immunosuppressive agents (cyclosporin, methotrexate, and mycophenolic acid)
* Vaccination of PPSV-23 (receiving childhood pneumococcal vaccination during infancy is eligible for this study)
* Pregnancy

Enrollment will be delayed 2 weeks for those subjects that can be included but have upper respiratory infection or viral illness to allow for natural resolution.

Ages: 19 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in asthma Control Status | approximately 1 year
  Change in asthma control status will be assessed at end of 1 year follow up. Included would be Asthma Control Test (ACT) Score

SECONDARY OUTCOMES:
Comparison of PPSV23 vaccine serotype specific antibody response between asthmatic and non-asthmatic smokers | Vaccine response will be measured at 4 to 6 weeks after administration of vaccine
  Vaccine response in form of serotype titers to pneumococcal antigens will be measured 4-6 weeks after vaccination and post vaccine titers will be compared with pre-vaccine titers between asthmatics and non-asthmatics (smokers)

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Divekar, MBBS, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No